CLINICAL TRIAL: NCT03881696
Title: Omalizumab as Monotherapy and as Adjunct Therapy to Multi-Allergen Oral Immunotherapy (OIT) in Food Allergic Children and Adults (CoFAR-11)
Brief Title: Omalizumab as Monotherapy and as Adjunct Therapy to Multi-Allergen OIT in Food Allergic Participants
Acronym: OUtMATCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry); Novartis Pharmaceuticals (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT CoFAR-11; CoFAR-11 (Other: Consortium for Food Allergy Research); NIAID CRMS ID#: 38625 (Other: DAIT NIAID)
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Peanut Allergy; Multi-food Allergy
Keywords: peanut allergic; multi-food allergic; omalizumab; placebo; multi-allergen oral immunotherapy (OIT); double-blind placebo-controlled food challenge (DBPCFC); oral food challenge (OFC)
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Stage 1:Omalizumab as Monotherapy (Experimental): Eligible participants are randomized to receive omalizumab by subcutaneous injection either every 2 weeks or every 4 weeks for 16 to 20 weeks. The dose administered and the dosing interval are determined by serum total IgE level and body weight (measured before the start of treatment) per the study drug dosing table.
  After 16 weeks of treatment, each participant will complete double-blind placebo-controlled food challenge (DBPCFCs) to each of their three specific foods to a cumulative dose of 6044 mg protein of each food.
  Throughout Stage 1, each participant will be instructed to strictly avoid all foods to which they are allergic.
  The first 60 participants who complete all four DBPCFCs at the end of Stage 1 will participate in the Stage 1 Open Label Extension (OLE).All other participants who complete all four DBPCFCs will move Stage 2 of the study.
  Interventions: Drug: Omalizumab
- Stage 1: Omalizumab OLE (Experimental): OLE: Open Label Extension, Long-Term Treatment with Omalizumab. Participants will receive 24 weeks of open label omalizumab in accordance with the omalizumab dosing table defined in the study protocol. Omalizumab is administered by subcutaneous injection either every 2 weeks or every 4 weeks for 24 weeks. The dose administered and the dosing interval are determined by serum total IgE level and body weight (measured before the start of treatment) per the study drug dosing table.
  After 24 weeks of treatment, each participant will complete DBPCFCs to each of their three specific foods to a cumulative dose of 8044 mg protein of each food. Each participant who completes all four DBPCFCs at the end of the Stage 1 OLE will move on to Stage 3 of the study.
  Throughout Stage 1 OLE, each participant will be instructed to strictly avoid all foods to which they are allergic.
  Interventions: Drug: Omalizumab
- Stage 1: Placebo for Omalizumab as Monotherapy (Placebo Comparator): Eligible participants are randomized to receive placebo for omalizumab by subcutaneous injection either every 2 weeks or every 4 weeks for 16 to 20 weeks. The dose administered and the dosing interval are determined by serum total IgE level and body weight (measured before the start of treatment) per the study drug dosing table.
  After 16 weeks of treatment, each participant will complete DBPCFCs to each of their three specific foods to a cumulative dose of 6044 mg protein of each food.
  Throughout Stage 1, each participant will be instructed to strictly avoid all foods to which they are allergic.
  The first 60 participants who complete all four DBPCFCs at the end of Stage 1 will participate in the Stage 1 OLE. All other participants who complete all four DBPCFCs will move Stage 2 of the study.
  Interventions: Drug: Placebo for Omalizumab
- Stage 2: Omalizumab (Experimental): Participants will receive eight weeks of treatment with open label omalizumab in accordance with the omalizumab dosing table specified in the study protocol, administered by subcutaneous injection. The dose administered and the dosing interval are determined by serum total IgE level and body weight (measured before the start of treatment) per the study drug dosing table.
  After completion of eight weeks of open label omalizumab, participants will be randomized 1:1 to either:
  * Omalizumab-facilitated oral immunotherapy (OIT): Open label omalizumab + Multi-allergen OIT for eight weeks, followed by placebo for omalizumab + Multi-allergen OIT for 44 weeks OR
  * Omalizumab + placebo OIT: Open label omalizumab + placebo for Multi-allergen OIT for eight weeks, followed by omalizumab + placebo for Multi-allergen OIT for 44 weeks.
  Throughout Stage 2, each participant will be instructed to strictly avoid all foods to which they are allergic.
  Interventions: Drug: Omalizumab
- Stage 2: Omalizumab-Facilitated OIT (Experimental): OIT: oral immunotherapy-Omalizumab as Adjunct Therapy to Multi-Allergen Oral Immunotherapy
  Participants randomized to open label omalizumab + Multi-allergen OIT for eight weeks, followed by placebo for omalizumab + Multi-allergen OIT for 44 weeks.
  Throughout Stage 2, each participant will be instructed to strictly avoid all foods to which they are allergic.
  Interventions: Drug: Omalizumab; Drug: Multi-Allergen Oral Immunotherapy
- Stage 2: Omalizumab + Placebo OIT (Experimental): OIT: oral immunotherapy Participants randomized to open label omalizumab + placebo for Multi-allergen OIT for eight weeks, followed by omalizumab + placebo for Multi-allergen OIT for 44 weeks.
  Throughout Stage 2, each participant will be instructed to strictly avoid all foods to which they are allergic.
  Interventions: Drug: Omalizumab; Drug: Placebo for Multi-Allergen Oral Immunotherapy
- Stage 3: DBPCFC Based Treatment (Other): DBPCFC Based Treatment-Long-term Follow-up Treatment Plan for Peanut and Each of the Two Other Participant-Specific Foods.
  Upon completion of the DBPCFCs at the end of Stage 1 OLE or Stage 2, each participant will receive a separate treatment plan for peanut and each of the two other participant-specific foods based on the results of the DBPCFCs. A treatment plan will include instructions for one of the following:
  * Long-term follow-up with dietary consumption of a food;
  * Long-term follow-up with avoidance of a food; or
  * Rescue OIT for a food.
  The treatment plan for each food may change throughout Stage 3 depending on a participant's response to treatment. Once a participant enters Stage 3, the participant will have a minimum of 12 months follow-up until at least December 2022.
  Note: Participants will be instructed to strictly avoid a food if they receive rescue OIT for the food during Stage 3.
  Interventions: Other: Double-Blind Placebo-Controlled Food Challenge Based Treatment

INTERVENTIONS:
Drug: Omalizumab — Omalizumab will be supplied in pre-filled syringes (PFS). PFS of omalizumab will be provided to the clinical research units as 75 mg and 150 mg dosage forms.
  Other Names: Xolair®
  Arms: Stage 1: Omalizumab OLE; Stage 1:Omalizumab as Monotherapy; Stage 2: Omalizumab; Stage 2: Omalizumab + Placebo OIT; Stage 2: Omalizumab-Facilitated OIT
Drug: Placebo for Omalizumab — Placebo contains the same ingredients as the omalizumab formulation, excluding omalizumab. Placebo will be supplied in pre-filled syringes (PFS). PFS of placebo will be provided to the clinical research units as 75 mg and 150 mg dosage forms.
  Other Names: Placebo
  Arms: Stage 1: Placebo for Omalizumab as Monotherapy
Drug: Multi-Allergen Oral Immunotherapy — Multi-allergen OIT will be any of the following drug products: peanut, milk, egg, wheat, cashew, hazelnut, and walnut (all food protein flours).
  A prescription for each participant for the appropriate dose of each of the allergens will be prepared. The pharmacist will compound the appropriate allergens and dispense the Multi-allergen OIT dose in a blinded (masked) fashion. The Clinical Research Unit (CRU) staff will administer food flour to the participant orally in an age-appropriate food vehicle (e.g., applesauce, pudding, etc.). Dosage will be administered according to the study protocol.
  Other Names: Multi-Allergen OIT
  Arms: Stage 2: Omalizumab-Facilitated OIT
Drug: Placebo for Multi-Allergen Oral Immunotherapy — Oat flour will be used for placebo for Multi-allergen OIT. Route: by mouth/oral. Dosage will be administered according to the study protocol.
  Other Names: Placebo for Multi-Allergen OIT
  Arms: Stage 2: Omalizumab + Placebo OIT
Other: Double-Blind Placebo-Controlled Food Challenge Based Treatment — Each participant will receive a separate treatment plan for peanut and each of the two other participant-specific foods. A treatment plan will include instructions for one of the following:
  * Long-term follow-up with dietary consumption of a food; or
  * Long-term follow-up with avoidance of a food; or
  * Rescue OIT for a food. The treatment plan for each food may change depending on a participant's response to prescribed treatment over time.
  Other Names: DBPCFC Based Treatment
  Arms: Stage 3: DBPCFC Based Treatment

SUMMARY:
This study is a multi-center, randomized, double-blind, placebo-controlled study in participants 1 to less than 56 years of age who are allergic to peanut and at least two other foods (including milk, egg, wheat, cashew, hazelnut, or walnut). While each participant may be allergic to more than two other foods, the primary endpoint/outcome in this study will only be assessed in peanut and two other foods for each participant. The primary objective of the study is to compare the ability to consume foods without dose-limiting symptoms during a double-blind placebo-controlled food challenge (DBPCFC), after treatment with either omalizumab or placebo for omalizumab.

DETAILED DESCRIPTION:
Food allergy affects about 15 million people in the United States. This includes 6 million children. The current treatment for food allergy is to avoid eating the foods that may cause an allergic reaction and have medications such as epinephrine (adrenaline) in case of a reaction. However, accidental exposures can be extremely difficult to avoid, particularly if you are allergic to multiple foods. The risks of accidental exposures and life-threatening reactions can place a large burden on patients and their families.

Investigators in this study would like to learn if omalizumab injections alone or in combination with multi-allergen oral immunotherapy (OIT) will help people with multiple food allergies eat foods to which they are allergic. Oral means that you will take the food allergen (peanut and 2 other foods to which you are allergic) by mouth. If you are allergic to more than 3 foods, this study will only provide OIT for peanut and 2 other foods.

There are 3 stages to the study:

In Stage 1, investigators would like to learn:

• If omalizumab stops or decreases allergic reactions to peanut and other common food allergens after taking it for a length of time.

Stage 1 will also have an extra part so that 60 participants will receive omalizumab and everyone (the investigators conducting the research and study participants) will know it. This is why it is called the open label extension. This part of the study will assist investigators in learning if receiving omalizumab for a longer time may work better at decreasing allergic reactions.

In Stage 2, investigators would like to learn:

• How a short course of omalizumab combined with Multi-allergen OIT compares with a longer course of omalizumab in decreasing allergic reactions.

In Stage 3, investigators would like to learn:

• If, after participants stop both treatments, will they be able to eat the peanut and the 2 other foods in the form that is normally eaten.

In all stages, investigators would like to learn:

* How safe and effective the treatments are and
* How the OIT affects the immune system.

Participation will last up to 56 months (4 years and 8 months).

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

1. Participant and/or parent/legal guardian must be able to understand and provide informed consent and/or assent, as applicable;
2. Peanut allergic: participant must meet all of the following criteria to minimize the chance that the participant will develop natural tolerance to peanut over the course of the study:

   1. Positive skin prick test (SPT) defined as ≥4 mm wheal greater than saline control) to peanut,
   2. Positive peanut immunoglobulin E (IgE), ≥6 kUA/L, at Screening or within three months of Screening, determined by ImmunoCap, and
   3. Positive double-blind placebo-controlled food challenge (DBPCFC), defined as experiencing dose-limiting symptoms at a single dose of ≤100 mg of peanut protein.
3. Allergic to at least two of the six other foods (milk, egg, wheat, cashew, hazelnut, walnut): each participant must meet all of the following criteria for at least two of the six other foods to minimize the chance that the participant will develop natural tolerance to at least two of the six other foods over the course of the study:

   1. Positive SPT (≥4 mm wheal) to food,
   2. Positive food specific IgE (≥6 kUA/L) at Screening or within three months of Screening, determined by ImmunoCap, and
   3. Positive DBPCFC, defined as experiencing dose-limiting symptoms at a single dose of ≤300 mg of food protein.
4. With body weight (as measured at Screening) and total serum IgE level (as measured within three months of Screening) suitable for omalizumab dosing;
5. If female of child-bearing potential, must have a negative urine or serum pregnancy test;
6. For women of childbearing potential, must agree to,during the treatment period and for 60 days after the last dose of study drug:

   * remain abstinent (refrain from heterosexual intercourse), or
   * use acceptable contraceptive methods (barrier methods, or
   * oral, injected, or implanted hormonal methods of contraception, or
   * other forms of hormonal contraception that have comparable efficacy).
7. Plan to remain in the study area of an OUtMATCH clinical research unit (CRU) during the trial; and
8. Be willing to be trained on the proper use of an epinephrine autoinjector for the duration of the study.

Exclusion Criteria:

Individuals who meet any of the following criteria are not eligible for enrollment as study participants:

1. Inability or unwillingness of a participant and/or parent/legal guardian to give written informed consent and/or assent or comply with the study protocol;
2. Clinically significant laboratory abnormalities at Screening;
3. Dose-limiting symptoms to the placebo portion of the Screening DBPCFC;
4. Sensitivity or suspected/known allergy to any ingredients (including excipients) of the

   * active or placebo oral food challenge (OFC) material,
   * multi-allergen oral immunotherapy (OIT), or
   * drugs related to omalizumab (e.g., monoclonal antibodies, polyclonal gamma globulin).

     * Note: Guidance for determination of sensitivity to excipients will be detailed in the study's Manual of Procedures (MOP).
5. Poorly controlled atopic dermatitis (AD) at Screening, per the Principal Investigator's PI's) discretion;
6. Poorly controlled or severe asthma/wheezing at Screening, defined by at least one of the following criteria:

   1. Global Initiative for Asthma (GINA) criteria regarding asthma control latest guidelines,
   2. History of two or more systemic corticosteroid courses within six months of Screening or one course of systemic corticosteroids within three months of Screening to treat asthma/wheezing,
   3. Prior intubation/mechanical ventilation for asthma/wheezing,
   4. One hospitalization or Emergency Department (ED) visit for asthma/wheezing within six months of Screening,
   5. Forced expiratory volume in one second (FEV1) <80 percent of predicted or FEV1/forced vital capacity (FVC) <75 percent, with or without controller medications (only for participants who are aged seven years or older and are able to perform spirometry), or
   6. Inhaled corticosteroid (ICS) dosing of >500 mcg daily fluticasone (or equivalent ICS based on the National Institutes of Health, National Heart, Lung, and Blood Institute (NHLBI) dosing chart).
7. History of severe anaphylaxis to participant-specific foods that will be used in this study, defined as neurological compromise or requiring intubation;
8. Treatment with a burst of oral, intramuscular (IM), or intravenous (IV) steroids of more than two days for an indication other than asthma/wheezing within 30 days of Screening;
9. Currently receiving oral, intramuscular, or intravenous corticosteroids, tricyclic antidepressants, or beta-blockers (oral or topical);
10. Past or current history of eosinophilic gastrointestinal (GI) disease within three years of Screening;
11. Past or current history of cancer, or currently being investigated for possible cancer;
12. Previous adverse reaction to omalizumab;
13. Past or current history of any immunotherapy to any of the foods being treated in this study (e.g., OIT, sublingual immunotherapy [SLIT], EPIT) within 6 months of Screening;
14. Treatment with monoclonal antibody therapy, such as omalizumab (Xolair®), dupilumab (Dupixent®), benralizumab (Fasenra™), mepolizumab (Nucala®), reslizumab (Cinqair®), or other immunomodulatory therapy within six months of Screening;
15. Currently on "build-up phase" of inhalant allergen immunotherapy (i.e., has not reached maintenance dosing). Note: Individuals tolerating maintenance allergen immunotherapy can be enrolled;
16. Inability to discontinue antihistamines for the minimum wash-out periods required for SPTs,or OFCs;
17. Current participation in another therapeutic or interventional clinical trial or participation within 90 days of Screening;
18. Use of investigational drugs within 24 weeks of Screening;
19. Pregnant or breastfeeding, or intending to become pregnant during the study or within 60 days after the last dose of omalizumab or placebo for omalizumab;
20. Has a first-degree relative already enrolled in the study; or
21. Past or current medical problems (e.g., severe latex allergy), history of other chronic diseases (other than asthma/wheezing, AD, or rhinitis) requiring therapy (e.g., heart disease, diabetes), findings from physical assessment, or abnormalities in clinical laboratory testing that are not listed above, which, in the opinion of the PI, may:

    * pose additional risks from participation in the study,
    * may interfere with the participant's ability to comply with study requirements, or
    * may impact the quality or interpretation of the data obtained from the study.

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 471 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2025-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Wood, MD, Study Chair — Department of Pediatrics at the Johns Hopkins University School of Medicine; Sharon Chinthrajah, MD, Study Chair — Department of Medicine, Stanford University School of Medicine
Locations (10):
- United States (10):
  - Arkansas Children's Hospital Research Institute: Department of Pediatrics, Allergy & Immunology, Little Rock, Arkansas
  - Stanford School of Medicine: Sean N. Parker Center for Allergy & Asthma Research, Stanford, California
  - National Jewish Health: Division of Pediatric Allergy and Clinical Immunology, Denver, Colorado
  - Emory University School of Medicine: Children's Healthcare of Atlanta Pediatrics, Atlanta, Georgia
  - Johns Hopkins Children's Center: Department of Allergy & Immunology, Baltimore, Maryland
  - Massachusetts General Hospital, Department of Medicine: Allergy & Clinical Immunology Unit, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai: Department of Pediatrics Allergy & Immunology, New York, New York
  - North Carolina Children's Hospital: Department of Pediatrics, Division of Allergy, Immunology and Rheumatology, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia: Division of Allergy and Immunology, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center: Division of Allergy and Immunology, Dallas, Texas

REFERENCES:
- [Background] Sampson HA, Berin MC, Plaut M, Sicherer SH, Jones S, Burks AW, Lindblad R, Leung DYM, Wood RA. The Consortium for Food Allergy Research (CoFAR): The first generation. J Allergy Clin Immunol. 2019 Feb;143(2):486-493. doi: 10.1016/j.jaci.2018.12.989. Epub 2018 Dec 23. PMID 30586557
- [Result] Wood RA, Togias A, Sicherer SH, Shreffler WG, Kim EH, Jones SM, Leung DYM, Vickery BP, Bird JA, Spergel JM, Iqbal A, Olsson J, Ligueros-Saylan M, Uddin A, Calatroni A, Huckabee CM, Rogers NH, Yovetich N, Dantzer J, Mudd K, Wang J, Groetch M, Pyle D, Keet CA, Kulis M, Sindher SB, Long A, Scurlock AM, Lanser BJ, Lee T, Parrish C, Brown-Whitehorn T, Spergel AKR, Veri M, Hamrah SD, Brittain E, Poyser J, Wheatley LM, Chinthrajah RS. Omalizumab for the Treatment of Multiple Food Allergies. N Engl J Med. 2024 Mar 7;390(10):889-899. doi: 10.1056/NEJMoa2312382. Epub 2024 Feb 25. PMID 38407394
- See also: Division of Allergy, Immunology, and Transplantation — http://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases — http://www.niaid.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was open from July 2019 through March 2023.
Pre-assignment Details: 471 Participants were enrolled during the recruitment period. 289 of the participants that enrolled did not meet the required eligibility criteria and therefore were considered trial screen failures. 180 participants went on to randomize in Stage 1. 2 participants met eligibility criteria after Stage 1 was completed and randomized directly into Stage 2.
Groups:
- Omalizumab: Omalizumab
- Placebo for Omalizumab: Placebo for Omalizumab
Period: Overall Study
Arm/Group | Omalizumab | Placebo for Omalizumab
Started | 120 | 60
Completed | 114 | 60
Not Completed | 6 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Subject withdrawal by parent or guardian | 1 | 0
Not completed — Failure to meet continuation criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set - Stage 1 (FA-S1): All participants who have been randomized to receive either omalizumab or placebo for omalizumab in Stage 1. Participants will be analyzed according to the treatment arm to which they were randomized in Stage 1, regardless of the treatment actually received in Stage 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo for Omalizumab | Total
Number analyzed (Participants) | 120 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (4.87) | 8.0 (5.19) | 7.8 (4.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 28 | 77
  Male | 71 | 32 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 14
  Not Hispanic or Latino | 110 | 56 | 166
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 12 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 4 | 14
  White | 74 | 37 | 111
  More than one race | 23 | 7 | 30
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 120 | 60 | 180
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] — Body Mass Index (kg/m²)
  kg/m² | 17.457 (3.0438) | 17.215 (3.6763) | 17.377 (3.2599)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by Stage 1 Treatment Assignment, Omalizumab Versus Placebo, Who Successfully Consume a Single Dose of ≥600 mg of Peanut Protein Without Dose-Limiting Symptoms During the DBPCFC Conducted at the End of Treatment Stage 1
Description: Number of participants who successfully consume a single dose of ≥600 mg of peanut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Population: Pediatric Full Analysis Set - Stage 1 (PFA-S1): All participants aged less than 18 years at randomization who have been randomized to either omalizumab or placebo for omalizumab in Stage 1. Participants will be analyzed according to the treatment arm to which they were randomized in Stage 1, regardless of the treatment actually received in Stage 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab | Placebo for Omalizumab
Number analyzed (Participants) | 118 | 59
Participants
  Success | 79 | 4
  Failure | 39 | 55
Statistical Analysis 1: Comparison: Omalizumab vs Placebo for Omalizumab; The null hypothesis is that the odds of 'success' (defined as consumption of a single dose of ≥600 mg of peanut protein without dose-limiting symptoms during the DBPCFC at the end of Stage 1) in omalizumab and placebo for omalizumab arms are equal. Participants missing the blinded OFC to peanut at the end of Stage 1 will be considered a 'failure' for the primary efficacy endpoint; Test type: Superiority; p < 0.00001, Fisher Exact — The a priori threshold for statistical significance was p < 0.0001 at the interim analysis OR p < 0.05 at the final analysis. Gatekeeping and multiple testing strategies were performed to ensure the overall family-wise error rate was ≤ 5%; Odds Ratio (OR) = 27.853, 95% CI 2-sided [9.1274 to 111.2144] — The odds ratio (OR) represents the odds of success among subjects randomized to omalizumab (numerator) compared to the odds of success among subjects randomized to placebo (denominator, reference group)

2. Secondary Outcome: Number of Participants by Stage 1 Treatment Assignment, Omalizumab Versus Placebo, Who Successfully Consume a Single Dose of ≥1000 mg of Cashew Protein Without Dose-limiting Symptoms During the DBPCFC Conducted at the End of Stage 1
Description: Number of participants who successfully consume a single dose of ≥1000 mg of cashew protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants by Stage 1 Treatment Assignment, Omalizumab Versus Placebo, Who Successfully Consume a Single Dose of ≥1000 mg of Milk Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 1
Description: Number of participants who successfully consume a single dose of ≥1000 mg of milk protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants by Stage 1 Treatment Assignment, Omalizumab Versus Placebo, Who Successfully Consume a Single Dose of ≥1000 mg of Egg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 1
Description: Number of participants who successfully consume a single dose of ≥1000 mg of egg protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

5. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Milk Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of milk protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

6. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Egg Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of egg protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

7. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Wheat Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of wheat protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

8. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Cashew Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of cashew protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

9. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Hazelnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of hazelnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

10. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Walnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of walnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

11. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Food Protein Without Dose-limiting Symptoms for at Least Two Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC), at the End of Stage 1
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of food protein without dose-limiting symptoms for at least two treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

12. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Food Protein Without Dose-limiting Symptoms for at Least Three Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC), at the End of Stage
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of food protein without dose-limiting symptoms for all three treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Peanut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1.
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of peanut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

14. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Wheat Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1.
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of wheat protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

15. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Hazelnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1.
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of hazelnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

16. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Walnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1.
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of walnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

17. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Food Protein Without Dose-limiting Symptoms for at Least Two Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of food protein without dose-limiting symptoms for at least two treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

18. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000mg of Food Protein Without Dose-limiting Symptoms for All Three Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume a single dose of ≥1000mg of food protein without dose-limiting symptoms for all three treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

19. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Peanut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of peanut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

20. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Milk Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of milk protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

21. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Egg Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of egg protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

22. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Wheat Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of wheat protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

23. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Cashew Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of cashew protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

24. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Hazelnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of hazelnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

25. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Walnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of walnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

26. Secondary Outcome: Proportion of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Food Protein Without Dose-limiting Symptoms for at Least Two Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of food protein without dose-limiting symptoms for at least two treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

27. Secondary Outcome: Proportion of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Food Protein Without Dose-limiting Symptoms for All Three Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC), at the End of Stage 1
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of food protein without dose-limiting symptoms for all three treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

28. Secondary Outcome: Proportion of Participants Who Successfully Consume 2 Doses of 2000 mg of Peanut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume 2 doses of 2000 mg of peanut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation]
Reporting Status: Not Posted

29. Secondary Outcome: Proportion of Participants Who Successfully Consume 2 Doses of 2000 mg of Milk Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume 2 doses of 2000 mg of milk protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

30. Secondary Outcome: Number of Participants Who Successfully Consume 2 Doses of 2000 mg of Egg Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume 2 doses of 2000 mg of egg protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

31. Secondary Outcome: Number of Participants Who Successfully Consume 2 Doses of 2000 mg of Wheat Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume 2 doses of 2000 mg of wheat protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

32. Secondary Outcome: Number of Participants Who Successfully Consume 2 Doses of 2000 mg of Cashew Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume 2 doses of 2000 mg of cashew protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

33. Secondary Outcome: Number of Participants Who Successfully Consume 2 Doses of 2000 mg of Hazelnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume 2 doses of 2000 mg of hazelnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

34. Secondary Outcome: Number of Participants Who Successfully Consume 2 Doses of 2000 mg of Walnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume 2 doses of 2000 mg of walnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

35. Secondary Outcome: Number of Participants Who Successfully Consume 2 Doses of 2000 mg of Food Protein Without Dose-limiting Symptoms for at Least Two Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume 2 doses of 2000 mg of food protein without dose-limiting symptoms for at least two treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

36. Secondary Outcome: Number of Participants Who Successfully Consume 2 Doses of 2000 mg of Food Protein Without Dose-limiting Symptoms for All Three Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 1
Description: Proportion of participants who successfully consume 2 doses of 2000 mg of food protein without dose-limiting symptoms for all three treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

37. Secondary Outcome: Number of Foods Consumed at a Single Dose of ≥600 mg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 1.
Description: Proportion of participants that were able to consume 0, 1, 2, or 3 foods at a threshold of ≥ 600 mg food protein during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

38. Secondary Outcome: Number of Foods Consumed at a Single Dose of ≥1000 mg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 1.
Description: Proportion of participants that were able to consume 0, 1, 2, or 3 foods at a threshold of ≥ 1000 mg food protein during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

39. Secondary Outcome: Number of Foods Consumed at ≥1 Dose of 2000 mg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 1
Description: Proportion of participants that were able to consume 0, 1, 2, or 3 foods at a threshold ≥ 1 dose of 2000 mg food protein during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

40. Secondary Outcome: Number of Foods Consumed at 2 Doses of 2000 mg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 1.
Description: Proportion of participants that were able to consume 0, 1, 2, or 3 foods at a threshold of 2 doses of 2000 mg food protein during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 1 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab or placebo for omalizumab. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 1: 16 to 20 weeks after Stage 1 treatment initiation
Reporting Status: Not Posted

41. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Peanut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of peanut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

42. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Milk Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of milk protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

43. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Egg Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of egg protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

44. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Wheat Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of wheat protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

45. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Cashew Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of cashew protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

46. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Hazelnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of hazelnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

47. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Walnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of walnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

48. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Food Protein Without Dose-limiting Symptoms for at Least Two Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of food protein without dose-limiting symptoms for at least two treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

49. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥600 mg of Food Protein Without Dose-limiting Symptoms for All Three Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥600 mg of food protein without dose-limiting symptoms for all three treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

50. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Peanut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of peanut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

51. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Milk Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of milk protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage treatment initiation
Reporting Status: Not Posted

52. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Egg Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of egg protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

53. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Wheat Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of wheat protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

54. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Cashew Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of cashew protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

55. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Hazelnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of hazelnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

56. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Walnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of walnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

57. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000 mg of Food Protein Without Dose-limiting Symptoms for at Least Two Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥1000 mg of food protein without dose-limiting symptoms for at least two treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

58. Secondary Outcome: Number of Participants Who Successfully Consume a Single Dose of ≥1000mg of Food Protein Without Dose-limiting Symptoms for All Three Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume a single dose of ≥1000mg of food protein without dose-limiting symptoms for all three treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

59. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Peanut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of peanut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

60. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Milk Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of milk protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

61. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000mg of Egg Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of egg protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

62. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000mg of Wheat Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥1 dose of 2000mg of wheat protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

63. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000mg of Cashew Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥1 dose of 2000mg of cashew protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

64. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Hazelnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of hazelnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

65. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Walnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of walnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

66. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Food Protein Without Dose-limiting Symptoms for at Least Two Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of food protein without dose-limiting symptoms for at least two treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

67. Secondary Outcome: Number of Participants Who Successfully Consume ≥1 Dose of 2000 mg of Food Protein Without Dose-limiting Symptoms for All Three Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥1 dose of 2000 mg of food protein without dose-limiting symptoms for all three treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

68. Secondary Outcome: Number of Participants Who Successfully Consume ≥2 Doses of 2000 mg of Peanut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥2 doses of 2000 mg of peanut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

69. Secondary Outcome: Number of Participants Who Successfully Consume ≥2 Doses of 2000 mg of Milk Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥2 doses of 2000 mg of milk protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

70. Secondary Outcome: Number of Participants Who Successfully Consume ≥2 Doses of 2000 mg of Egg Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥2 doses of 2000 mg of egg protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

71. Secondary Outcome: Number of Participants Who Successfully Consume ≥2 Doses of 2000 mg of Wheat Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥2 doses of 2000 mg of wheat protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

72. Secondary Outcome: Number of Participants Who Successfully Consume ≥2 Doses of 2000 mg of Cashew Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) Conducted in a Controlled Clinic Setting, at the End of Stage 2
Description: Proportion of participants who successfully consume ≥2 doses of 2000 mg of cashew protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

73. Secondary Outcome: Number of Participants Who Successfully Consume ≥2 Doses of 2000 mg of Hazelnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥2 doses of 2000 mg of hazelnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

74. Secondary Outcome: Number of Participants Who Successfully Consume ≥2 Doses of 2000 mg of Walnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥2 doses of 2000 mg of walnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

75. Secondary Outcome: Number of Participants Who Successfully Consume ≥2 Doses of 2000 mg of Food Protein Without Dose-limiting Symptoms for at Least Two Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume ≥2 doses of 2000 mg of food protein without dose-limiting symptoms for at least two treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

76. Secondary Outcome: Number of Participants Who Successfully Consume ≥2 Doses of 2000 mg of Food Protein Without Dose-limiting Symptoms for All Three Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage
Description: Proportion of participants who successfully consume ≥2 doses of 2000 mg of food protein without dose-limiting symptoms for all three treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

77. Secondary Outcome: Number of Participants Who Successfully Consume 3 Doses of 2000 mg of Peanut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume 3 doses of 2000 mg of peanut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

78. Secondary Outcome: Number of Participants Who Successfully Consume 3 Doses of 2000 mg of Milk Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume 3 doses of 2000 mg of milk protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

79. Secondary Outcome: Number of Participants Who Successfully Consume 3 Doses of 2000 mg of Egg Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume 3 doses of 2000 mg of egg protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

80. Secondary Outcome: Proportion of Participants Who Successfully Consume 3 Doses of 2000 mg of Wheat Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume 3 doses of 2000 mg of wheat protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

81. Secondary Outcome: Number of Participants Who Successfully Consume 3 Doses of 2000 mg of Cashew Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume 3 doses of 2000 mg of cashew protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

82. Secondary Outcome: Number of Participants Who Successfully Consume 3 Doses of 2000 mg of Hazelnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume 3 doses of 2000 mg of hazelnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

83. Secondary Outcome: Number of Participants Who Successfully Consume 3 Doses of 2000 mg of Walnut Protein Without Dose-limiting Symptoms During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume 3 doses of 2000 mg of walnut protein without dose-limiting symptoms during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

84. Secondary Outcome: Number of Participants Who Successfully Consume 3 Doses of 2000 mg of Food Protein Without Dose-limiting Symptoms for at Least Two Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume 3 doses of 2000 mg of food protein without dose-limiting symptoms for at least two treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

85. Secondary Outcome: Number of Participants Who Successfully Consume 3 Doses of 2000 mg of Food Protein Without Dose-limiting Symptoms for All Three Treated Food Allergens During the Double-blind Placebo-controlled Oral Food Challenge (DBPCFC) at the End of Stage 2
Description: Proportion of participants who successfully consume 3 doses of 2000 mg of food protein without dose-limiting symptoms for all three treated food allergens during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

86. Secondary Outcome: Number of Foods Consumed at a Single Dose of ≥600 mg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 2.
Description: Proportion of participants that were able to consume 0, 1, 2, or 3 foods at a threshold of ≥ 600 mg food protein during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

87. Secondary Outcome: Number of Foods Consumed at a Single Dose of ≥1000 mg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 2.
Description: Proportion of participants that were able to consume 0, 1, 2, or 3 foods at a threshold of ≥ 1000 mg food protein during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

88. Secondary Outcome: Number of Foods Consumed at ≥1 Dose of 2000 mg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 2.
Description: Proportion of participants that were able to consume 0, 1, 2, or 3 foods at a threshold of ≥ 1 dose of 2000 mg food protein during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

89. Secondary Outcome: Number of Foods Consumed at ≥2 Doses of 2000 mg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 2.
Description: Proportion of participants that were able to consume 0, 1, 2, or 3 foods at a threshold of 2 doses of 2000 mg food protein during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

90. Secondary Outcome: Number of Foods Consumed at 3 Doses of 2000 mg Protein Without Dose-limiting Symptoms During the DBPCFC at the End of Stage 2.
Description: Proportion of participants that were able to consume 0, 1, 2, or 3 foods at a threshold of 3 doses of 2000 mg food protein during the double-blind placebo-controlled oral food challenge (DBPCFC) conducted in a controlled clinic setting, at the end of Stage 2 treatment, to compare the ability of participants to consume foods without dose-limiting symptoms during a DBPCFC after treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT. Dose-limiting symptoms are those that in the view of the principal investigator indicate a true allergic reaction.
Time Frame: During the DBPCFC at the end of Stage 2: 60 to 64 Weeks after Stage 2 treatment initiation
Reporting Status: Not Posted

91. Secondary Outcome: During Stage 1: Occurrence of Adverse Event(s) Related to Study Therapy Regimen, Omalizumab Versus Placebo
Description: To evaluate safety during treatment with either omalizumab or placebo for omalizumab during Stage 1 masked (blinded) treatment.
Time Frame: Up to 20 Weeks after initiating Stage 1 randomized treatment initiation
Reporting Status: Not Posted

92. Secondary Outcome: During Stage 1 OLE : Occurrence of Adverse Event(s) Related Study to Therapy Regimen, Open Label Extension (OLE)
Description: To evaluate safety during this open label omalizumab study therapy regimen during Stage 1.
Time Frame: Up to 28 Weeks after initiating Stage 1 Open Label omalizumab study therapy regimen
Reporting Status: Not Posted

93. Secondary Outcome: During Stage 2: Occurrence of Adverse Event(s) Related to Study Therapy Regimen
Description: To evaluate safety during treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT during Stage 2.
Time Frame: Up to 64 Weeks after initiating Stage 2 study therapy regimen
Reporting Status: Not Posted

94. Secondary Outcome: During Stage 3: Occurrence of Adverse Event(s) Related to Oral Food Intake
Description: To evaluate safety after the conclusion of treatment with either omalizumab-facilitated oral immunotherapy (OIT) or omalizumab + placebo OIT during a follow-up period in which participants either received guided dietary instructions and/or rescue OIT for up to three foods (Stage 3).
Time Frame: Up to 2 years after initiating Stage 3 Oral Food Intake regimen
Reporting Status: Not Posted

95. Secondary Outcome: Number of Weeks in Each Eight-week Period During Stage 3 Where ≥300 mg Protein of Each Food is Consumed at Least Twice Per Week
Description: To compare dietary consumption of foods after the conclusion of treatment with either omalizumab facilitated OIT or omalizumab + placebo OIT during a follow-up period in which participants either received guided dietary instructions and/or rescue oral immunotherapy (OIT) for up to three foods (Stage 3).
Time Frame: From initial 8-week period during Stage 3 up to the last possible 8-week period during Stage 3 (i.e., Up to N=13 possible 8-week intervals during a 2-year period of time in Stage 3)
Reporting Status: Not Posted

96. Secondary Outcome: Number of Weeks in Each Eight-week Period During Stage 3 Where Each Food is Not Consumed
Description: as for outcome 95
Time Frame: as for outcome 95
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Stage 1 treatment-emergent AEs were collected from first administration of study drug through end of Stage 1 (up to 20 weeks) or early termination from the study.
Description: Treatment-emergent AEs for all 180 participants that randomized into Stage 1. Reporting does not include the OLE period.
Arm/Group | Omalizumab | Placebo for Omalizumab
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/60
Serious Adverse Events (participants affected / at risk) | 4/120 | 1/60
Other Adverse Events (participants affected / at risk) | 62/120 | 37/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (N=120) | Placebo for Omalizumab (N=60)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (N=120) | Placebo for Omalizumab (N=60)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Injection site reaction (General disorders) | 11 (20) | 5 (6)
Pyrexia (General disorders) | 7 (7) | 2 (2)
Hypersensitivity (Immune system disorders) | 25 (34) | 23 (34)
Corona virus infection (Infections and infestations) | 8 (8) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (4)
Influenza (Infections and infestations) | 3 (3) | 3 (4)
Nasopharyngitis (Infections and infestations) | 3 (4) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (8) | 3 (3)
Viral infection (Infections and infestations) | 5 (6) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT03881696/Prot_003.pdf
  • Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT03881696/SAP_004.pdf
  • Informed Consent Form (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03881696/ICF_005.pdf